CLINICAL TRIAL: NCT00091728
Title: Hormonal Contraception, Cervical Ectopy, and STDs
Brief Title: Hormonal Contraception and Risk of Chlamydia and Gonorrhea
Status: Terminated | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: HD7034
Record Dates: First submitted 2004-09-16; First posted 2004-09-20 (Estimated); Last update posted 2005-11-07 (Estimated); Status verified 2004-09

CONDITIONS: Chlamydia Infection; Neisseriaceae Infection
Keywords: epidemiology; relative risk; cervical ectopy; hormonal contraceptives; sexually transmitted infections
MeSH Terms: conditions — Chlamydia Infections; Neisseriaceae Infections; Sexually Transmitted Diseases | interventions — Medroxyprogesterone Acetate; Contraceptives, Oral, Combined

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: Depo Medroxyprogesterone acetate
Drug: Combined oral contraceptives

SUMMARY:
There are biological reasons to suspect that hormones may affect the risk of a woman becoming infected with a sexually transmitted disease. The evidence on this issue to date is mixed and previous studies have methodologic flaws making it difficult to draw conclusions about the results.

This study compares the risk of developing either Chlamydial or Gonorrheal infection among three groups of women: those using combined oral contraceptives (birth control pills); those using the injectable hormone (brand name Depo Provera); and those women using non-hormonal contraceptive methods.

DETAILED DESCRIPTION:
The study was designed to examine the relationship between hormonal contraceptive use and possible increased risk of Chlamydial and Gonococcal sexually transmitted infections, and to determine if any increased risk appeared to be mediated by the extent of cervical ectopy.

Eight hundred and nineteen women, ages 15 to 45 years, were recruited from an inner city clinic and from a nearby suburban clinic. The women were classified into three groups based on type of contraceptive used. One group used oral contraceptives; the second used injectable depo-medroxyprogesterone acetate (DMPA); and the third group used non-hormonal contraceptive methods. Women from each group were followed at 3, 6, and 12 months after enrollment to determine if a new infection with Chlamydia or Gonorrhea had occurred and to evaluate the extent of cervical ectopy present.

ELIGIBILITY:
Inclusion Criteria:

* Female age 15 to 45 years
* no hormone use at enrollment
* not pregnant or planning pregnancy

Exclusion Criteria:

* Cervical cancer presently or in history
* hysterectomy, cone biopsy, or cervical cryotherapy

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1200
Dates: Start 1997-09; Study Completion 2001-08

CONTACTS AND LOCATIONS:
Overall Officials: Charles Morrison, Ph.D., Principal Investigator — Family Health International, RTP, N.C.; Paul Blumenthal, M.D., Principal Investigator — Maryland Planned Parenthood